CLINICAL TRIAL: NCT00655499
Title: An Open-label Phase II Trial of Panitumumab Plus Irinotecan for Patients With Advanced Metastatic Colorectal Cancer Without KRAS Mutation (Wild-type) in Third-line Chemotherapy (FOLFOX/XELOX ± Bevacizumab and Irinotecan Alone or FOLFIRI/CAPIRI ± Bevacizumab)
Brief Title: Panitumumab and Irinotecan as Third-Line Therapy in Treating Patients With Metastatic Colorectal Cancer
Acronym: PIMABI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000593012; GERCOR-PIMABI-C07-1 (Other: GERCOR); 2007-004806-28 (EudraCT Number); EU-20836 (Other: EU Clinical Trials Register); AMGEN-GERCOR-PIMABI-C07-1 (Other: GERCOR, AMGEN)
Record Dates: First submitted 2008-04-09; First posted 2008-04-10 (Estimated); Results first posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2016-08

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; adenocarcinoma of the rectum; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer; recurrent colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Panitumumab; Irinotecan; In Situ Hybridization; In Situ Hybridization, Fluorescence; Gene Expression Profiling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab + CPT11 (irinotecan hydrochloride) (Experimental): 1 cycle every 14 days (J1= J15)
  Interventions: Drug: Panitumumab; Drug: Irinotecan hydrochloride; Genetic: Chromogenic in situ hybridization; Genetic: Fluorescence in situ hybridization; Genetic: Gene expression analysis; Other: Laboratory biomarker analysis

INTERVENTIONS:
Drug: Panitumumab — 6 mg/kg
  Other Names: Vectibix
Drug: Irinotecan hydrochloride — 180 mg/kg
  Other Names: Camptosar
Genetic: Chromogenic in situ hybridization
Genetic: Fluorescence in situ hybridization
Genetic: Gene expression analysis
Other: Laboratory biomarker analysis

SUMMARY:
RATIONALE: Monoclonal antibodies, such as panitumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving panitumumab together with irinotecan may kill more tumor cells.

PURPOSE: This phase II clinical trial is studying giving panitumumab together with irinotecan to see how well it works as third-line therapy in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the objective response rate when panitumumab is administered in combination with irinotecan hydrochloride as third-line therapy in patients with advanced metastatic colorectal cancer without KRAS mutation (wild type) previously treated with FOLFOX or XELOX chemotherapy with or without bevacizumab and irinotecan hydrochloride alone or FOLFIRI or CAPIRI chemotherapy with or without bevacizumab.

Secondary

* To assess the efficacy in terms of disease control rate, duration of response, time to response, progression-free survival, time to progression, time to treatment failure, and duration of stable disease.
* To assess the efficacy and safety of this regimen, followed by panitumumab alone in patients who discontinue third-line irinotecan hydrochloride due to toxicity.

Tertiary

* To correlate this regimen with EGFR expression, detection of the functional genetic polymorphisms of the EGFR gene, EGFR gene amplification (FISH), EGFR activation detection, EGFR downstream protein and gene expression parameters, proteomics, and epigenetics.

OUTLINE: This is a multicenter study.

Patients receive panitumumab IV over 30-90 minutes and irinotecan hydrochloride IV over 90 minutes on day 1. Patients who discontinue irinotecan hydrochloride may receive panitumumab monotherapy. Courses repeat every 14 days in the absence of disease progression and unacceptable toxicity.

Archived tumor tissue specimens are obtained at baseline for correlative laboratory studies. Tissue samples are analyzed for EGFR amplification status by chromogenic in situ hybridization and fluorescence in situ hybridization, KRAS and KRAF mutations, and STAT3 expression.

After completion of study therapy, patients are followed at approximately 56 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal adenocarcinoma

  * Metastatic disease
* Wild-type KRAS (no mutation) by allelic discrimination on tumor DNA
* Measurable disease (≥ 10 mm) per modified RECIST criteria
* Previously treated for metastatic disease with oxaliplatin and fluoropyrimidines (i.e., fluorouracil/folinic acid or capecitabine) with or without bevacizumab, and irinotecan hydrochloride alone or in combination with fluoropyrimidines (i.e., fluorouracil/folinic acid or capecitabine) with or without bevacizumab
* Must have paraffin-embedded tissue or unstained tumor slides from primary or metastatic tumor available for correlative studies
* Must be registered with a national health care system (CMU included)
* No CNS metastases unless previously treated or asymptomatic, provided patient has been off steroids for at least 30 days prior to study treatment

PATIENT CHARACTERISTICS:

* WHO performance status of 0-2
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Creatinine < 150 μmol/L or creatinine clearance > 30 mL/min
* AST ≤ 3 times upper limit of normal (ULN) (5 times ULN if liver metastases present)
* ALT ≤ 3 times ULN (5 times ULN if liver metastases present)
* Bilirubin ≤ 1.5 times ULN
* Magnesium normal
* No significant cardiovascular disease, including unstable angina or myocardial infarction within the past 6 months
* No history of treated or untreated ventricular arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double barrier contraception during and for 6 months after completion of study treatment
* No other malignant tumors within the past five years except basocellular carcinoma, in situ cancer of the cervix or uterus, or any UDAW cancers for which there has been complete resection for at least three years
* No known hypersensitivity to an excipient (vehicle) of panitumumab or known hypersensitivity of irinotecan trihydrate chlorhydrate or known hypersensitivity excipient (vehicle) of irinotecan hydrochloride
* No history of interstitial pneumonitis, pulmonary fibrosis or evidence of interstitial pneumonitis, or pulmonary fibrosis on baseline chest CT scan
* No active inflammatory bowel disease, other bowel disease causing chronic diarrhea (defined as > 4 loose stools per day), or bowel occlusion
* No history of Gilbert syndrome
* No history of any medical condition that may increase the risks associated with study participation or may interfere with the interpretation of the study results
* No known positive test for HIV infection, hepatitis C virus, chronic active hepatitis B infection
* No comorbid disease that would increase risk of toxicity
* No disorder that would compromise the patient's ability to give written informed consent and/or comply with study procedures
* Must be willing and able to comply with study requirements
* No grade IV toxicity associated with a past treatment with irinotecan hydrochloride

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 14 days since prior treatment for systemic infection
* No prior or concurrent anti-EGFR antibody therapy (e.g., cetuximab) or treatment with small molecule EGFR tyrosine kinase inhibitors (e.g., erlotinib hydrochloride)

  * Patients who discontinued their first dose of anti-EGFR therapy (i.e., cetuximab) because of an infusion reaction are eligible
* More than 30 days since prior and no other concurrent investigational agent (no delay for non-investigational treatment)
* More than 14 days since prior CYP3A4 enzyme, including anticonvulsant medication (e.g., phenytoin, phenobarbital, or carbamazepine)
* More than 14 days since prior rifampicin
* More than 14 days since prior radiotherapy and recovered
* More than 7 days since prior and no concurrent ketoconazole
* More than 28 days since prior and no concurrent major surgical procedure
* Concurrent topical, oral, or IV antibiotics used to treat skin- or nail-related toxicities are allowed at the investigator's discretion
* No other concurrent experimental or approved anti-tumor therapies (e.g., bevacizumab), chemotherapy other than irinotecan hydrochloride, non-palliative radiotherapy, or systemic steroids (except when used for symptomatic skin or nail-related toxicities requiring withholding of the panitumumab dose, as chemotherapy premedication, or for an infusion reaction)
* No concurrent St. John's wort (i.e., Hypericum perforatum)
* No concurrent phenobarbital, clarithromycin, erythromycin, HIV protease inhibitors, cyclosporine or tacrolimus, or nefazodone
* Concurrent minor surgery, procedures, or surgery arising as needed or necessary allowed
* Concurrent elective surgery allowed in patients eligible for surgical resection of metastases as curative therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Andre, MD, Principal Investigator — GERCOR - Multidisciplinary Oncology Cooperative Group
Locations (9):
- France (9):
  - Centre Paul Papin, Angers
  - Hopital Prive Jean Mermoz, Lyon
  - Hopital Clinique Claude Bernard, Metz
  - Centre Hospitalier Intercommunal Le Raincy - Montfermeil, Montfermeil
  - Hopital Pitie-Salpetriere, Paris
  - Hopital Bichat - Claude Bernard, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - Hopital Foch, Suresnes

REFERENCES:
- [Derived] Andre T, Blons H, Mabro M, Chibaudel B, Bachet JB, Tournigand C, Bennamoun M, Artru P, Nguyen S, Ebenezer C, Aissat N, Cayre A, Penault-Llorca F, Laurent-Puig P, de Gramont A; GERCOR. Panitumumab combined with irinotecan for patients with KRAS wild-type metastatic colorectal cancer refractory to standard chemotherapy: a GERCOR efficacy, tolerance, and translational molecular study. Ann Oncol. 2013 Feb;24(2):412-419. doi: 10.1093/annonc/mds465. Epub 2012 Oct 5. PMID 23041588

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2008 to Oct. 2010, 69 patients were enrolled in the study, 4 were not eligible.The study was conducted in 11 French centers
Pre-assignment Details: Patient wih pathologically confirmed mCRC, KRAS codon 12 and 13 wild type, previously treated with irinotecan, oxaliplatin, fluoropyrimidines and bevacizumab. Eligibility criteria also included : age ≥ 18 years, normal hematopoietic , hepatic and renal functions, measurable disease.No prior treatment with anti-EGFR antibodies.
Groups:
- Panitumumab Combined With Irinotecan: 65 patients were eligible (69 patients were enrolled and 4 patients were not eligible).
Period: Overall Study
Arm/Group | Panitumumab Combined With Irinotecan
Started | 69
Completed | 65
Not Completed | 4
Not completed — not eligible | 4

BASELINE CHARACTERISTICS:
Population: 69 patients were enrolled in the study. 4 patients were not eligible.Baseline measures are provided for 65 patients
Groups:
- Panitumumab Combined With Irinotecan: 1cycle every 14 days (J1=J15). Panitumumab : 6mg/kg in IV infusion over 60 minutes on day 1. Irinotecan : 180mg/m² in IV infusion over 90 minutes on day 1 just after panitumumab administration
Arm/Group | Panitumumab Combined With Irinotecan
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 31
Age, Continuous [Mean (Full Range); unit: years] | 62 [34 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 39
Region of Enrollment [Number; unit: participants]
  France | 65
ECOG Performance status [Number; unit: participants] — The ECOG Performance Status is a method to assess the functional status of a patient.
  * ECOG - PS 0 : Fully active, able to carry on all pre-disease performance without restriction
  * ECOG - PS 1 : Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  * ECOG - PS 2 :Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  participants
    ECOG performance status - PS = 0 | 25
    ECOG - PS=1 | 33
    ECOG - PS=2 | 7
Primary tumor type [Number; unit: participants]
  Colon | 45
  Rectum | 17
  Both | 3
Number of metastatic sites [Number; unit: participants]
  1 metastatic site | 37
  >1 metastatic site | 28
Adjuvant chemotherapy [Number; unit: participants]
  Yes | 17
  No | 48
Time between diagnosis and inclusion [Number; unit: participants]
  < 12 months | 13
  ≥12-24 months | 21
  > 24 months | 31
First line chemotherapy [Number; unit: participants]
  Oxaliplatin-based therapy | 42
  Irinotecan-based therapy | 22
  Oxaliplatin- and irinotecan-based therapy | 1
Second line chemotherapy [Number; unit: participants]
  Oxaliplatin-based therapy | 14
  Irinotecan-based therapy | 43
  No second line | 8
Prior treatment with bevacizumab [Number; unit: participants]
  No | 12
  Yes | 53

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) During the Combination Therapy Phase
Description: Per the modified Response Evaluation Criteria in Solid Tumors (m-RECIST) for target lesions and radiogically assessed (CT Scans; optionally MRI): Complete Response (CR; Disappearance of all target lesions) or Partial Response (PR; At least a 30% decrease in the sum of the LD of target lesions) during the combination therapy phase.Overall Response (OR) = CR + PR.
Time Frame: Up to 20 months
Population: Panitumumab combined with irinotecan
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Panitumumab Combined With Irinotecan: 69 patients were enrolled in the study. 4 patients were not eligible. 65 eligible patients were analysed
Arm/Group | Panitumumab Combined With Irinotecan
Number analyzed (Participants) | 65
percentage of patients
  Whole study population | 29.2 [18.2 to 40.3]
  Confirmed wild-type KRAS population: number analyzed (Participants) | 54
  Confirmed wild-type KRAS population | 35.2 [22.4 to 47.9]
  All wild-type population: number analyzed (Participants) | 41
  All wild-type population | 46.3 [31.1 to 61.6]
  Patients with KRAS, NRAS or BRAF mutations: number analyzed (Participants) | 19
  Patients with KRAS, NRAS or BRAF mutations | 0 [0 to 0]

2. Secondary Outcome: Disease Control Rate (DCR)
Description: Per the modified Response Evaluation Criteria in Solid Tumors (m-RECIST) for target lesions and radiogically assessed (CT Scans; optionally MRI): confirmed complete (CR; Disappearance of all target lesions) or partial response (PR; At least a 30% decrease in the sum of the longest diameter of target lesions), or stable disease (SD; Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression, taking as reference the nadir longest diameter since the treatment started) while on the combination therapy treatment phase or over the entire treatment strategy. DCR = CR / PR / SD
Time Frame: Up to 20 months
Population: Panitumumab combined with irinotecan
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panitumumab Combined With Irinotecan
Number analyzed (Participants) | 65
percentage of participants
  Overall period | 63.1 [51.3 to 74.8]
  Confirmed wild-type KRAS population: number analyzed (Participants) | 54
  Confirmed wild-type KRAS population | 66.7 [54.1 to 79.2]
  All Wild-type population: number analyzed (Participants) | 41
  All Wild-type population | 80.5 [68.3 to 92.6]
  Patients with KRAS, NRAS or BRAF mutation: number analyzed (Participants) | 19
  Patients with KRAS, NRAS or BRAF mutation | 21.1 [2.72 to 39.4]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as time from enrollment date to date of first radiologically observed progression or death (whichever comes first) during the combination therapy phase or over the entire treatment strategy.
  Per the Response Evaluation Criteria in Solid Tumors (RECIST) analyzed using Kaplan-Meier methods and the quartiles and event rates at various weeks presented with 95% CIs.
Time Frame: Up to 20 months
Population: Panitumumab combined with irinotecan
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panitumumab Combined With Irinotecan
Number analyzed (Participants) | 65
percentage of participants
  Overall Period | 5.5 [3.7 to 7.6]
  Confirmed wild-type KRAS population: number analyzed (Participants) | 54
  Confirmed wild-type KRAS population | 6.3 [3.7 to 8.7]
  All wild-type population: number analyzed (Participants) | 41
  All wild-type population | 8.7 [5.5 to 10.4]
  Patient with KRAS, NRAS or BRAF mutations: number analyzed (Participants) | 19
  Patient with KRAS, NRAS or BRAF mutations | 1.9 [1.5 to 2.4]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as time from inclusion to death (from any cause or to the last date the patient was known to be alive) during the combination therapy phase or over the entire treatment strategy.
  Per the Response Evaluation Criteria in Solid Tumors (RECIST) analyzed using Kaplan-Meier methods and the quartiles and event rates at various weeks presented with 95% CIs.
Time Frame: Up to 20 months
Population: Panitumumab combined with irinotecan
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Panitumumab Combined With Irinotecan
Number analyzed (Participants) | 65
percentage of participant
  Study population | 9.7 [6.6 to 15.8]
  Confirmed wild-type KRAS population: number analyzed (Participants) | 54
  Confirmed wild-type KRAS population | 11.9 [6.8 to 18.2]
  All wild-type population: number analyzed (Participants) | 41
  All wild-type population | 15.8 [9.5 to 25.1]
  Patients with KRAS, NRAS or BRAF mutation: number analyzed (Participants) | 19
  Patients with KRAS, NRAS or BRAF mutation | 4.6 [3.3 to 7.9]

ADVERSE EVENTS:
Time Frame: From the date of inclusion to 56 ± 3 days after the last dosing of study treatment
Description: Adverse events (AE) were collected during the treatment period and safety follow-up phases and were graded using NCI-CTCAE version 3.0.
Groups:
- Panitumumab + CPT11: 1 cycle every 14 days (J1= J15)
  panitumumab: Panitumumab : 6mg/kg
  irinotecan hydrochloride: 180mg/kg
  chromogenic in situ hybridization
  fluorescence in situ hybridization
  gene expression analysis
  laboratory biomarker analysis
Arm/Group | Panitumumab + CPT11
Serious Adverse Events (participants affected / at risk) | 10/65
Other Adverse Events (participants affected / at risk) | 29/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panitumumab + CPT11 (N=65)
Occular hemorraghe (Vascular disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
General physical health deterioration (General disorders) | 3 (3)
occlusion (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab + CPT11 (N=65)
skin toxicity (Skin and subcutaneous tissue disorders) | 21 — grade 3/4
Neutropenia (Blood and lymphatic system disorders) | 8 — grade 3/4
Diarrhoea (Gastrointestinal disorders) | 10 — grade 3/4
Mucositis (Gastrointestinal disorders) | 1 — grade 3/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No